CLINICAL TRIAL: NCT05848271
Title: A Patient Registry and Natural History Study of Patients with Biallelic HPDL Mutations
Brief Title: Natural History Study of Patients with HPDL Mutations
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: New York University (Other); Universität Tübingen (Other); Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Joseph Gleeson, professor, neuroscience, University of California, San Diego
Other Study IDs: HPDL_NHS_001
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Mitochondrial Encephalomyopathies; Hereditary Spastic Paraplegia; Spastic Paraplegia; White Matter Disease; Neonatal Encephalopathy; Mutation; Genetic Disease
Keywords: HPDL; HPDL related neonatal mitochondrial encephalopathy; HPDL related hereditary spastic paraplegia; Spastic paraplegia-83; Neurodevelopmental disorder with progressive spasticity and brain white matter abnormalities
MeSH Terms: conditions — Mitochondrial Encephalomyopathies; Spastic Paraplegia, Hereditary; Paraplegia; Leukoencephalopathies; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — dry blood spots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HPDL deficiency: Patients with HPDL mutations
  Interventions: Other: Patient Registry; Other: Dry blood spots sampling

INTERVENTIONS:
Other: Patient Registry — Participants who have been diagnosed with HPDL mutations will be enrolled to patient registry.
Other: Dry blood spots sampling — Dry blood splots require 500nl of blood.

SUMMARY:
This study uses medical records that allow retrospective data extraction of clinical manifestation to assess the natural history of HPDL mutations

DETAILED DESCRIPTION:
A novel mitochondrial disease arises from mutations in HPDL, which codes for 4-hydroxyphenylpyruvate dioxygenase-like protein. The main purpose of this study is to establish a patient registry to gather medical data from consenting HPDL mutation patients worldwide. From longitudinal data, we will be able to figure out the natural history of the disease, and genotype-phenotype correlation. Dry blood spots will be collected to develop biomarkers to understand the disease better.

ELIGIBILITY:
Inclusion Criteria:

* Any individuals diagnosed with HPDL variants
* Clinical diagnosis can include:

  * HPDL-related hereditary spastic paraplegia (HSP)
  * HPDL-related neonatal mitochondrial encephalopathy
  * Spastic paraplegia -83 (SPG83)
  * Neurodevelopmental disorder with progressive spasticity and brain white matter abnormalities (NEDSWMA)

Exclusion Criteria:

* Any known genetic abnormality (other than HPDL mutation)
* Any condition that, in the opinion of the Site Investigator, could put the participant at undue risk and/or would ultimately prevent the completion of study procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The gene HPDL has been linked to an infantile neurodegenerative condition. The affected patients have various clinical manifestations from spastic paraplegia to NEDSWMA. Severely affected patients exhibit developmental delay, seizures, and spasticity, and can lead to death.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinician questionnaire | 12 months
  Clinician-reported clinical and genetic confirmation of HPDL mutations

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Gleeson, Principal Investigator — UCSD
Locations (1):
- Eun Hae Lee, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghosh SG, Lee S, Fabunan R, Chai G, Zaki MS, Abdel-Salam G, Sultan T, Ben-Omran T, Alvi JR, McEvoy-Venneri J, Stanley V, Patel A, Ross D, Ding J, Jain M, Pan D, Lubbert P, Kammerer B, Wiedemann N, Verhoeven-Duif NM, Jans JJ, Murphy D, Toosi MB, Ashrafzadeh F, Imannezhad S, Karimiani EG, Ibrahim K, Waters ER, Maroofian R, Gleeson JG. Biallelic variants in HPDL, encoding 4-hydroxyphenylpyruvate dioxygenase-like protein, lead to an infantile neurodegenerative condition. Genet Med. 2021 Mar;23(3):524-533. doi: 10.1038/s41436-020-01010-y. Epub 2020 Nov 14. PMID 33188300
- [Background] Banh RS, Kim ES, Spillier Q, Biancur DE, Yamamoto K, Sohn ASW, Shi G, Jones DR, Kimmelman AC, Pacold ME. The polar oxy-metabolome reveals the 4-hydroxymandelate CoQ10 synthesis pathway. Nature. 2021 Sep;597(7876):420-425. doi: 10.1038/s41586-021-03865-w. Epub 2021 Sep 1. PMID 34471290
- [Derived] Lee EH, Kim-Mcmanus O, Yang JH, Haas R, Zaki MS, Abdel-Salam GMH, Nakamura Y, Abdel-Hamind MS, Ebrahimi-Fakhari D, Alecu JE, Brunetti-Pierri N, Srinivasan VM, Gowda VK, Gross S, Alanay Y, Najarzadeh Totbati P, Yadavilli M, Friedman L, Ojeda NM, Gleeson JG. HPDL Variant Type Correlates With Clinical Disease Onset and Severity. Ann Clin Transl Neurol. 2025 Jul;12(7):1360-1367. doi: 10.1002/acn3.70047. Epub 2025 May 14. PMID 40368591
- See also: website for patient registration — http://neurosciences.ucsd.edu/research/labs/gleeson/hpdl/index.html